CLINICAL TRIAL: NCT02099851
Title: Endovascular Carotid Body Ablation in Patients With Treatment- Resistant Hypertension: A Safety and Feasibility Study.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Noblewell (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL1003-CIBIEM
Record Dates: First submitted 2014-03-26; First posted 2014-03-31 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Carotid body ablation (Experimental): Patients undergoing the unilateral endovascular ablation of the right or left carotid body.
  Interventions: Device: Carotid body ablation (Cibiem)

INTERVENTIONS:
Device: Carotid body ablation (Cibiem)
  Other Names: Cibiem Carotid Body Modulation System

SUMMARY:
This is a prospective, observational, multicenter trial to evaluate the safety and feasibility of selective endovascular unilateral carotid body ablation in patients with treatment-resistant hypertension. All patients will be followed for two (2) years following treatment.

DETAILED DESCRIPTION:
The investigators propose a new method of treatment, unilateral carotid body ablation, for treatment- resistant hypertensive patients to restore more normal blood pressure control, which will reduce cardiovascular morbidity and mortality in these patients. This strategy will increase the number of therapeutic options available to many patients and their physicians as well as offering the potential of normal blood pressure to those patients in whom blood pressure remains elevated despite vigorous, drug or device based therapies.

ELIGIBILITY:
Inclusion Criteria:

* Age of participants will be 18-75 years.
* Treatment-resistant hypertensive subjects on medical management.
* Office systolic blood pressure (oBP) ≥ 160mmHg.
* Daytime mean ambulatory BP (ABPM) ≥ 140 mmHg.
* Persistent hypertension on at least three anti-hypertensive medications, including a diuretic, at stable, maximum tolerated dose within the last 90 days.
* No evidence for causes of secondary HTN (hypertension ) following thorough clinical assessment.
* At least one carotid body detected in CT angiography of the neck, defined as an hyper-enhanced ovoid structure strongly located poster-medially from the area of carotid bifurcation.
* Ability to give and giving informed consent to participate in the study.
* Women of child-bearing potential have a negative pregnancy test.

Exclusion Criteria:

* Calculated GFR (glomerular filtration rate) < 30ml/min/m2
* Obstructive carotid atherosclerotic disease which precludes safe delivery of ablation catheter or performance of ablation
* Must be at least 6 months post renal denervation therapy.
* Oxygen saturation at rest below 92%.
* Requirement for oxygen therapy to maintain oxygen saturation.
* Severe untreated obstructive sleep apnea (defined as an apnea-hypopnea index (AHI) ≥ 30/hour during Polysomnography associated with an average minimum oxygen desaturation of < 85%.
* Patients wish to participate in mountain climbing, sky diving or free diving.
* Pregnancy or anticipation of pregnancy.
* Acute coronary syndrome or unstable angina < 6 months before scheduled procedure.
* History of repeated episodes of hypoglycemia with hypoglycemic unawareness.
* Known diabetic autonomic neuropathy.
* History of, or current atrial fibrillation (AF).
* Life expectancy of less than 24 months due to other disease.
* Intravenous or inhaled recreational drug use.
* Excessive use of alcohol or sedatives (alcohol intake > 28 units/week).
* Morbid obesity (BMI >40).
* Febrile illness within two weeks of participation.
* History of Stroke, transient ischaemic attack (TIA) or significant chronic neurological condition in medical history.
* History of spontaneous intracranial hemorrhage within past 12 months.
* Unable to tolerate exposure to the radiopaque contrast agent.
* Unable to tolerate aspirin and/or other anti-coagulation; anti-platelet medication.
* Femoral arterial access is not possible.
* Presence of carotid artery dissection prior to the index procedure.
* Atherosclerotic disease involving vessels adjoining the carotid body, marked vessel tortuosity or other anatomical findings that preclude safe placement of the guiding catheter or the investigational system, and the delivery of RF energy.
* Carotid body is not within reach of the investigational system due to position within the carotid bifurcation or distance of the CB (carotid body) from the femoral access point.
* Other abnormal angiographic findings that indicate the patient is at risk of a stroke, such as carotid or intracranial aneurysm, arteriovenous malformation (AVM), other developmental or traumatic vascular lesion or tumor.
* Dementia or confusion precluding the patient's full understanding of the information required for informed consent and full participation in the study.
* Unable to attend schedule follow up appointments at one (1)_month, three (3) months, six (6) months, one (1) year and two (2) years post treatment.
* History of gastrointestinal bleeding within the last six (6) months.
* Active or treated malignancies in the last twelve (12) months.
* Patient is participating in another clinical study for which follow-up is currently on going.
* Patient with non-cardiac co-morbidities and life expectancy < 2 year.
* Patient has a condition that, in the opinion of the Investigator, precludes participation, including willingness to comply with all follow-up procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-03; Primary Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 3 months
  Safety and feasibility of selective endovascular unilateral carotid body ablation in patients with treatment-resistant hypertension employing a radiofrequency catheter designed specifically for this indication.

SECONDARY OUTCOMES:
Change of Blood Pressure | 3 months
  Change from Baseline Blood Pressure at 3 months

CONTACTS AND LOCATIONS:
Locations (2):
- Na Homolce Hospital, Roentgenova 2, Prague, Czechia
- Department of Hypertension and Diabetology, Medical University of Gdansk, Gdansk, Poland